CLINICAL TRIAL: NCT03947970
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Metabolism of [14C] CR845 in Patients With End Stage Renal Disease on Hemodialysis and in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics and Metabolism of [14C] CR845 (Difelikefalin) in Patients With End Stage Renal Disease on Hemodialysis and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR845-100302
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Hemodialysis; Healthy
Keywords: Hemodialysis; Difelikefalin; Dialysis; CR845; CKD; ESRD (end stage renal disease)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] CR845 (Experimental): Subjects will receive a single dose of [14C] CR845 IV solution administered as an IV bolus on Day 1.
  Interventions: Drug: [14C] CR845

INTERVENTIONS:
Drug: [14C] CR845 — Subjects will receive a single dose of 230 mcg CR845 solution containing 100 microcuries [14C] CR845, administered via IV bolus (the total dose of CR845 will range from 1.7 to 3.1 mcg/kg)

SUMMARY:
The objectives of this study are to evaluate the in vivo metabolite profiling and characterization of CR845 administered intravenously (IV) in patients on hemodialysis (HD) and in healthy subjects; and to determine the pharmacokinetics of radiolabeled [14C] CR845 administered as a single IV bolus in patients on HD and in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-radiolabeled dose, non-randomized study in 6 male patients on HD and 6 healthy male subjects. The study will consist of a Screening Period, a Study Period, and an End-of-Study assessment.

ELIGIBILITY:
Key Inclusion Criteria for Healthy Subjects

* Body mass index (BMI) within the range of 18 to 30 kg/m2, inclusive, and body weight not less than 75 kg;
* Vital signs at Screening must be within the following ranges and stable (measured in sitting position after at least 5 minutes' rest);

  * Systolic blood pressure (SBP) ≥100 and ≤140 mmHg;
  * Diastolic blood pressure (DBP) ≥50 and ≤90 mmHg;
  * Heart rate (HR) ≥50 and ≤100 beats per minute (bpm).
* Must be in good health as determined by past medical history, physical examination, ECG, vital sign assessments, and clinical laboratory tests at Screening. Any subjects with abnormalities noted at Screening or at any time before dosing on Day 1 must be approved by the Investigator and Medical Monitor.

Key Inclusion Criteria for patients on HD

* If taking concurrent medications, must be on a stable dose for at least 14 days prior to dosing and the dosing regimen should remain stable for the duration of the study;
* Prescription dry body weight of ≥75 kg and ≤135 kg at Screening;
* Must be receiving HD 3 times weekly and have been on dialysis for at least 3 months prior to Screening;
* For a minimum of 1 month before Day 1, must have stable controlled blood pressure that in the Investigator's opinion will not interfere with study conduct;
* Demonstrated adequate dialysis measurements (at least two Kt/V measurements ≥1.2 or two urea reduction ratio [URR] measurements ≥65%) during the 3 months prior to Screening

Key Exclusion Criteria:

* Has a concomitant disease or any medical condition that, in the opinion of the Investigator, could pose undue risk to the patient, impede completion of the study procedures, or would compromise the validity of the study measurements, including, but not limited to:

  * Known or suspected history of alcohol, narcotic, or other drug abuse, or substance dependence within 12 months prior to Screening;
  * Significant systolic or diastolic heart failure (eg, New York Heart Association Class IV congestive heart failure [Appendix 1]);
  * Severe mental illness or cognitive impairment (eg, dementia);
  * Any other relevant acute or chronic medical or neuropsychiatric condition.
* History of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator;
* Use of any beverages and foods containing alcohol, quinine (tonic water), grapefruit, broccoli, Brussels sprouts, Seville oranges, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to dosing with study medication without evaluation and approval by the Investigator;
* Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins, chapparal, comfrey, germander, gin bu huan, kava, pennyroyal, skullcap, St. John's Wort, or valerian) within 7 days prior to dosing with study medication;
* Use of any new prescription medication from 14 days prior to dosing with study medication without evaluation and approval by the Investigator;
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days prior to dosing with study medication, and that, in the Investigator's judgment, may impact subject safety or the validity of the study results;
* Positive results for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg);
* Is a healthy subject with positive results for hepatitis C virus (HCV) antibody at Screening. Note: Subjects with HD who test positive for HCV antibody may be allowed to enroll at the discretion of the Principal Investigator if their liver function tests are not otherwise clinically significant;
* Has donated blood or has had an acute loss of blood (˃500 mL) during the 3 months prior to study drug administration;
* Previous administration of any [14C] labeled drug substance within 1 year of study drug administration;
* Has irregular bowel habits. "Irregular" being defined for the purpose of this study as NOT having a bowel movement at least every 2 days.)
* Has been involved in an occupation that requires monitoring for radiation exposure (eg, X-ray technician);

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Measure of the [14C] CR845 and total radioactivity (total [14C] CR845-equivalents) in plasma, urine, feces, and dialysate will be determined. | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD
Extent of recovery of [14C] CR845 and radioactivity related to [14C] CR845 in plasma, urine, feces, and dialysate, as applicable, will be derived. | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD
Cumulative amount of [14C] CR845 and [14C] CR845-equivalents in urine and feces over the collection period will be calculated. | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD
Presence of possible CR845 metabolites will be assessed. | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD
Quantitation of possible CR845 metabolites will be assessed. | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD

SECONDARY OUTCOMES:
Frequency and severity of adverse events by treatment group | Day 1 to up to 7 days post dose in healthy volunteers and Day 1 to up to 14 days post dose in patients on HD

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (1):
- Cara Therapeutics Study Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stark JG, Noonan PK, Spencer RH, Bhaduri S, O'Connor SJ, Menzaghi F. Pharmacokinetics, Metabolism, and Excretion of Intravenous [14C]Difelikefalin in Healthy Subjects and Subjects on Hemodialysis. Clin Pharmacokinet. 2023 Sep;62(9):1231-1241. doi: 10.1007/s40262-023-01262-2. Epub 2023 Jun 28. PMID 37369955